CLINICAL TRIAL: NCT06017921
Title: Effect of Eszopiclone on Adherence to Continuous Positive Airway Pressure (CPAP) and Severity of Insomnia in Patients With Comorbidity Between Insomnia and Obstructive Sleep Apnea (COMISA)
Brief Title: Effect of Eszopiclone on Adherence to CPAP and Severity of Insomnia in Patients With COMISA
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Pedro Rodrigues Genta, Principal Investigador, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ComisaEszopiclone
Record Dates: First submitted 2023-05-10; First posted 2023-08-30 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Obstructive Sleep Apnea; Insomnia
Keywords: COMISA; Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Initiation and Maintenance Disorders | interventions — Eszopiclone

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eszopiclone (Active Comparator): Eszopiclone 3mg at bed time for 14 days
  Interventions: Drug: Eszopiclone 3 mg
- Placebo (Placebo Comparator): Placebo at bed time for 14 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eszopiclone 3 mg — Patients starting CPAP treatment will be randomized to either Eszopiclone or Placebo arm
  Arms: Eszopiclone
Drug: Placebo — Patients starting CPAP treatment will be randomized to either Eszopiclone or Placebo arm
  Arms: Placebo

SUMMARY:
The comorbidity between obstructive sleep apnea (OSA) and insomnia (COMISA) is common, and associated with poorer sleep quality. CPAP adherence among COMISA patients is worst than among those with OSA only. The investigators will compare the effect of Eszopiclone 3mg or placebo for 14 days on adherence to CPAP after 30 days and after 6 months.

DETAILED DESCRIPTION:
The comorbidity between OSA and insomnia (COMISA) is common. COMISA leads to additive impairment of quality of sleep and quality of life compared to patients with insomnia or OSA alone. Patients with COMISA demonstrate worse adherence to CPAP compared to patients with isolated OSA. The best therapeutic approach for patients with COMISA is still unclear. Hypnotics have not been tested among patients with COMISA and indication for CPAP.

The investigators will compare the effect of Eszopiclone 3mg or placebo for 14 days on adherence to CPAP after 30 days and after 6 months. In addition, the investigators will assess the effect eszopiclone on insomnia severity, quality of life, anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Insomnia;
* Moderate or severe OSA (AHI ≥ 15 events/h), diagnosed by polysomnography.

Exclusion Criteria:

* Craniofacial anatomical abnormalities or severe otorhinolaryngological disorders that potentially impair CPAP use;
* Use of hypnotics for more than 7 days in the last 2 months;
* Renal dysfunction (serum creatinine >2mg/dL);
* Severe liver or cardiac dysfunction;
* Alcoholism;
* Previous CPAP or mandibular advancement device for OSA treatment in the last 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-08-24 (Actual); Primary Completion 2025-03-20 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Short-term CPAP adherence (use > 4 hours per night through Resmed program) | 4 weeks
  Compare the effect of Eszopiclone 3mg or placebo for 14 days on one-month CPAP adherence (use > 4 hours per night through Resmed program) after 4 weeks days.
  Adherence to CPAP will be assess by the average number of hours of use (>=4h). The investigators will use Resmed's program for this analysis.

SECONDARY OUTCOMES:
Long-term CPAP adherence (use > 4 hours per night through Resmed program) Compare sleep quality, insomnia and anxiety | 6 months
  Compare the effect of Eszopiclone 3mg or placebo for 14 days on 6 months CPAP adherence (use > 4 hours per night through Resmed program), sleep quality, insomnia and anxiety through questionnaries.
  Adherence to CPAP will be assess by the average number of hours of use (>=4h). The investigators will use Resmed's program for this analysis.
  The sleep quality, insomnia and anxiety will be assess through questionnaires.

CONTACTS AND LOCATIONS:
Locations (1):
- Sleep Laboratory, Heart Institute, Pulmonary Division, Hospital das Clínicas da Universidade de São Paulo, São Paulo, Brazil